CLINICAL TRIAL: NCT05853510
Title: Are Mid-term Functional Outcomes Different in Unilateral and Bilateral Developmental Dysplasia of the Hip? A Cross-sectional Study
Brief Title: Mid-term Functional Comparisons of Unilateral and Bilateral Developmental Dysplasia of the Hip
Status: Completed | Type: Observational
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Raziye Şavkın, Associate Professor, Pamukkale University
Other Study IDs: 60116787-020-125130/20
Record Dates: First submitted 2023-05-02; First posted 2023-05-10 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Developmental Dysplasia of the Hip
MeSH Terms: conditions — Developmental Dysplasia of the Hip

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Unilateral developmental dysplasia of the hip: Diagnosed with developmental dysplasia of the hip and treated with a hip abduction brace in one hip.
- Bilateral developmental dysplasia of the hip: Diagnosed with developmental dysplasia of the hip and treated with a hip abduction brace in two hips.

SUMMARY:
The annual number of live births in Türkiye is 1,112,859 in 2020 and the estimated incidence of developmental dysplasia of the hip (DDH) is between 5 and 15 per 1000 live births. The implementation of the National DDH Early Diagnosis and Treatment Program by the Türkiye Republic of the Ministry of Health in 2010 significantly reduced the number of patients with DDH diagnosed more than 6 months later. If not appropriately treated, DDH can cause a decrease in the number of healthy life years, and workforce losses, which consequently burdens the social security system and government budget. The vast majority of clinical trials comprise risk factors associated with complications after treatment of DDH. Moreover, studies involving functional assessments are generally focused on adult DDH patients with surgical indications. To the best of the investigators' knowledge, mid-term patient-reported and performance-based functionality has not been examined in conservatively treated patients. In addition, it is not known whether the diagnosis of unilateral and bilateral DDH in these patients will make a difference in daily activities which require bilateral functionality of the lower limbs. Therefore, in this study, the investigators examined and compared the mid-term patient-reported and performance-based functional outcomes in patients with unilateral and bilateral DDH treated with a hip abduction brace. This study provides new data on mid-term functionality in children with unilateral and bilateral DDH. It can guide determining the lower extremity functional levels of school-age children with DDH, regular follow-up, early diagnosis, and treatment planning for problems.

DETAILED DESCRIPTION:
The annual number of live births in Türkiye is 1,112,859 in 2020 and the estimated incidence of developmental dysplasia of the hip (DDH) is between 5 and 15 per 1000 live births. The implementation of the National DDH Early Diagnosis and Treatment Program by the Türkiye Republic of the Ministry of Health in 2010 significantly reduced the number of patients with DDH diagnosed more than 6 months later. If not appropriately treated, DDH can cause a decrease in the number of healthy life years, and workforce losses, which consequently burdens the social security system and government budget. The vast majority of clinical trials comprise risk factors associated with complications after treatment of DDH. Moreover, studies involving functional assessments are generally focused on adult DDH patients with surgical indications. To the best of the investigators' knowledge, mid-term patient-reported and performance-based functionality has not been examined in conservatively treated patients. In addition, it is not known whether the diagnosis of unilateral and bilateral DDH in these patients will make a difference in Daily activities which require bilateral functionality of the lower limbs. Therefore, in this study, the investigators examined and compared the mid-term patient-reported and performance-based functional outcomes in patients with unilateral and bilateral DDH treated with a hip abduction brace. This study provides new data on mid-term functionality in children with unilateral and bilateral DDH. It can guide determining the lower extremity functional levels of school-age children with DDH, regular follow-up, early diagnosis, and treatment planning for problems.

The vast majority of clinical trials comprise risk factors associated with complications after treatment of DDH. Moreover, studies involving functional assessments are generally focused on adult DDH patients with surgical indications. To the best of the investigators' knowledge, mid-term patient-reported and performance-based functionality has not been examined in conservatively treated patients. In addition, it is not known whether the diagnosis of unilateral and bilateral DDH in these patients will make a difference in activities such as jumping rope, double-leg jumping, walking, and dynamic balance, which require bilateral functionality of the lower limbs. Therefore, the aim of this study is to examine and compare the mid-term patient-reported and performance-based functional outcomes in patients with unilateral and bilateral DDH treated with a hip abduction brace.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with developmental dysplasia of the hip and treated with a hip abduction brace

Exclusion Criteria:

* teratological hip dislocations,
* hip avascular necrosis,
* comorbid disease such as cerebral palsy, myelomeningocele, hypoxic encephalopathy, muscular dystrophy and leukoencephalopathy,
* receiving different treatments before.

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients who were treated with hip abduction brace in the orthopedics and traumatology department of a university hospital from January 2010 to January 2016 were screened from the hospital registry system. Eligible 72 patients were contacted by telephone and invited to participate in the present study and 54 patients agreed to participate. A total of 35 patients were able to complete all assessments and their data were analyzed. 16 patients had unilateral and 19 patients had bilateral developmental dysplasia of the hip.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2021-11-11 (Actual); Primary Completion 2022-02-11 (Actual); Study Completion 2022-09-11 (Actual)

PRIMARY OUTCOMES:
Radiographs | 2 hours
  Standard pelvic AP radiographs taken at the first and last admission of the patients were used for radiological evaluation. The acetabular index angle of Hilgenreiner and the centeredge angle of Wiberg were measured. The Tönnis radiographic classification was used for patients with ossified femoral head, and the IHDI classification was used for other patients.
Lower Extremity Functional Scale | 30 minutes
  Lower Extremity Functional Scale was used for assess functional status in musculoskeletal dysfunction affecting the lower extremities. The scale mainly consists of 20-items and is a 5-point Likert type (0 = extreme difficulty or or unable to perform activity and 4 = no difficulty). Total score ranged from 0 to 80 points, with higher scores indicating better functional status.
10 meters walking test | 10 minutes
  10 meters walking test was used for assessing the walking speed over a distance of 10 meters
Double-leg vertical jump test | 15 minutes
  The double-leg vertical jump test was used to determine the strength and functional characteristics of the lower extremity extensor muscles. Participants stood upright with feet positioned shoulder width apart, and hands at their hips (to reduce the impact of arm movement). Patients were instructed to jump as high as possible with both legs.
Jump rope | 10 minutes
  Jump rope assesses the strength of the lower extremity muscles. Patients were asked to jump rope for 60 seconds and the number of repetitions was recorded
STAR excursion balance test | 10 minutes
  STAR excursion balance test was used to measure dynamic balance in children. The test was performed with both extremities. In order to reduce the time required to perform the test, reach in 3 directions was measured anterior, posteromedial, and posterolateral, respectively. To normalize the distances reached, the reach distance was divided by the leg length and multiplied by 100.

CONTACTS AND LOCATIONS:
Overall Officials: Raziye Şavkın, Dr, Principal Investigator — Pamukkale University
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No